CLINICAL TRIAL: NCT01013597
Title: A Phase II Trial of LBH589 in Patients With Metastatic Medullary Thyroid Cancer and Radioactive Iodine Resistant Differentiated Thyroid Cancer
Brief Title: Trial of LBH589 in Metastatic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2009-0173; CO08322 (Other: University of Wisconsin Carbone Cancer Center); H-2009-0173 (Other: Institutional Review Board); NCI-2011-00715 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2009-10-28; First posted 2009-11-13 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2017-03

CONDITIONS: Thyroid Carcinoma
Keywords: thyroid; medullary; differentiated; radioiodine-resistant; LBH589; panobinostat
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — LBH589 20mg by mouth three times weekly (Monday/Wednesday/Friday) for 28-day cycles.
  Other Names: panobinostat

SUMMARY:
The purpose of this study is to evaluate the tumor response rate in patients with metastatic medullary thyroid cancer (MTC) or radioiodine resistant differentiated thyroid cancer (DTC) after receiving treatment with LBH589 20 mg by mouth, three times weekly. Time to progression, overall survival, toxicity, tolerability, and Notch1 protein expression patterns will also be evaluated.

DETAILED DESCRIPTION:
Medullary thyroid cancer (MTC) is a neuroendocrine tumor and accounts for 3-5% of cases of thyroid cancer. The majority of patients with MTC do not present with early stage disease. Differentiated thyroid cancer (DTC) accounts for >90% of all thyroid cancers. In a sub-set of patients, thyroid cells become resistant to I-131 radioiodine therapy and subsequently develop distant metastases. In both MTC and DTC, systemic chemotherapy for metastatic disease is largely ineffective.

LBH589 is a histone deacetylase (HDAC) with recently demonstrated activity to inhibit the Notch1 signaling pathway in MTC cancer cells and suppress tumor cell proliferation in DTC cancer cells. This clinical trial will evaluate the tumor response rate of LBH589 in patients with metastatic MTC or radioactive iodine resistant DTC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic medullary or differentiated thyroid cancer. Diagnosis must be confirmed at University of Wisconsin
* Patients must have measurable disease as defined by RECIST.
* At least 3 weeks from the completion of major surgery, chemotherapy, or other systemic therapy or local liver therapy to study registration
* No concurrent chemotherapy or radiation therapy
* ECOG Performance Status of ≤ 2
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Adequate bone marrow, kidney, liver function
* Left ventricular ejection fraction ≥ the lower limit of the institutional normal
* Those with differentiated thyroid cancer must have radioactive iodine resistant disease, defined by failure to incorporate 131-Iodine after therapy, FDG-avidity on a PET scan, or progression of measurable disease after 131-Iodine therapy or an allergy to radioactive iodine
* Hypertension must be well controlled (to less than 150/90 mmHg) on a stable regimen of anti-hypertensive therapy

Exclusion Criteria:

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
* Impaired cardiac function
* Concomitant use of drugs with a risk of causing torsades de pointes
* Patients with unresolved diarrhea > CTCAE grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
* Other concurrent severe and/or uncontrolled medical conditions
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after last study drug administration. Women of childbearing potential must have a negative serum pregnancy test within 7 days of the first administration of oral LBH589.
* Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment
* Patients with a history of another primary malignancy that, in the opinion of the investigator, would interfere with the assessment of the primary endpoints of the study
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Traynor, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - St. Vincent Regional Cancer Center CCOP, Green Bay, Wisconsin
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LBH589
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | LBH589
Number analyzed (Participants) | 13
Age, Customized [Number; unit: participants]
  30-39 years | 1
  40-49 years | 2
  50-59 years | 2
  60-69 years | 6
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate to LBH589.
Description: per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v.1.0) for target lesions and assessed by CT/MRI: "Response" includes Complete Response (CR, disappearance of all target lesions), or Partial Response (PR, >=30% decrease in the sum of the longest diameter of target lesions). "No Response" includes Stable Disease (SD, neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease), and Progressive Disease (PD, at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s).)
Time Frame: Every 8 weeks.
Measure: Number; unit: participants
Arm/Group | LBH589
Number analyzed (Participants) | 13
participants
  No response | 13
  Response | 0

2. Secondary Outcome: Protein Expression Patterns of Notch1 in Thyroid Tissue Samples.
Time Frame: End of study
Population: Notch1 protein expression was not measured due to lack of efficiency of study intervention
Arm/Group | LBH589
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Progression of Thyroid Cancer
Description: Progression is defined using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Time to progression is defined as the number of days from the day of first LBH589 administration to the day the patient experienced an event of disease progression or death, whichever came first. Progression was assessed every 3 months until death or up to 5 years, whichever occurred first.
Time Frame: Every 3 months until progression up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LBH589
Number analyzed (Participants) | 13
months | 3.6 [1.8 to 5.8]

4. Secondary Outcome: Overall Survival
Description: For a given patient, overall survival (OS) is defined as the number of days from the day of first LBH589 administration until the patient's death. If a patient was alive at the time of analysis, then the patient's data is censored at the date of the last available evaluation.Survival was assessed every three months until death or final data analysis, whichever occurred first.
Time Frame: Every 3 months up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LBH589
Number analyzed (Participants) | 13
months | 18.4 [5.8 to NA] — upper limit not reached

5. Secondary Outcome: Impact of LBH589 on Tumor Markers for Thyroid Cancer
Description: Change in serum Thyroglobulin level from baseline to end of treatment. Treatment continued until either extraordinary medical circumstances, disease progression, toxicity, subject withdrawal, or death. At the time subjects came off of study treatment for one of the reasons already listed, a sample was collected for tumor markers.
Time Frame: Baseline and end of treatment, up to 1 year
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LBH589
Number analyzed (Participants) | 11
ng/mL | 4.58 (716.65)
Statistical Analysis 1: Comparison: LBH589; Test type: Superiority or Other; p = 0.98, t-test, 2 sided

6. Secondary Outcome: Toxicity of LBH589
Description: Most frequent toxicities at least possibly related to panobinostat, grades 2-4 (grading based on NCI common terminology criteria for adverse events CTCAE version 3). Toxicities were collected from the time the patient provided informed consent until 4 weeks after the patient stopped LBH589.
Time Frame: Every 4 weeks, up to 5 years
Measure: Number; unit: participants
Arm/Group | LBH589
Number analyzed (Participants) | 13
participants
  Anemia | 3
  Leukopenia | 7
  Neutropenia | 7
  Lymphopenia | 8
  Thrombocytopenia | 8
  Hypoalbuminemia | 3
  Fatigue | 8
  Diarrhea | 4
  Headache | 1
  Bone Pain | 1
  Hyperglycemia | 1
  Hypocalcemia | 2
  Asthenia | 1
  Rash | 1
  Anorexia | 4
  Anxiety | 1
  Elevated GGT | 1
  Pulmonary embolism | 1

7. Secondary Outcome: Tolerability of LBH589
Description: Tolerability and toxicity were not assessed separately, therefore tolerability is reported as toxicity.
Time Frame: Every 4 weeks, up to 5 years
Arm/Group | LBH589
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | LBH589
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LBH589 (N=13)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Death, NOS (General disorders) | 3
Hemorrhage/bleeding (General disorders) | 1 — neck lesion
Colitis, infectious (Infections and infestations) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Other (Nervous system disorders) | 1 — Subdural hematoma after fall
Pleural effusion, non-malignant (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes